CLINICAL TRIAL: NCT06605703
Title: The Comparative Effectiveness of Step-down Treatment Options for Weight Management After Discontinuation of Semaglutide and Tirzepatide: A Randomized Controlled Trial (GLP1 Transition Trial)
Brief Title: A Randomized Controlled Trial Comparing the Effectiveness of Different Treatment Options for Weight Management After Discontinuation of Semaglutide and Tirzepatide (GLP1 Transition Trial)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: WW International Inc (Industry)
Responsible Party: Principal Investigator, Jamil Alkhaddo, Medical Director, Clinical Development, WW International Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLP1 Transition Trial
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- WW Clinic - No medications (Experimental): Participants in this group receive behavioral or lifestyle support from WW Clinic. They receive no medications.
  Interventions: Behavioral: WW Clinic
- WW Clinic + Meds v1 (Experimental): Participants in this group receive behavioral or lifestyle support from WW Clinic. They receive medications prescribed through WW Clinic.
  Interventions: Behavioral: WW Clinic; Drug: Bupropion-Naltrexone
- WW Clinic + Meds v2 (Experimental): Participants in this group receive behavioral or lifestyle support from WW Clinic. They receive medications prescribed through WW Clinic.
  Interventions: Behavioral: WW Clinic; Drug: Bupropion-Naltrexone-Metformin

INTERVENTIONS:
Behavioral: WW Clinic — Telehealth platform that specializes in medical weight management and integrates the behavioral and lifestyle support from WW.
Drug: Bupropion-Naltrexone — Bupropion-Naltrexone
  Arms: WW Clinic + Meds v1
Drug: Bupropion-Naltrexone-Metformin — Bupropion-Naltrexone-Metformin
  Arms: WW Clinic + Meds v2

SUMMARY:
The study compares the effectiveness of treatment options for weight management after discontinuing semaglutide and tirzepatide. The primary outcome is absolute and percentage weight change at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Previous hx of BMI of >30 or BMI of >27 with one or more weight related medically qualifying condition (hypertension, dyslipidemia, sleep apnea, cardiovascular disease)
* Currently taking Wegovy, Ozempic, Mounjaro or Zepbound and have been for at least 6 months
* At least 15% body weight loss since taking Wegovy, Ozempic, Mounjaro, or Zepbound
* Willing to stop taking their GLP-1 medication or is discontinuing due to circumstances such as access, cost, coverage, choice, or any other reason
* Ability to provide informed consent prior to any trial-related activities
* Able to read and write in English

Exclusion Criteria:

* BMI <22 kg/m2
* Diabetes
* Previous surgical obesity treatment
* Currently pregnant or intending to become pregnant during the study
* Breastfeeding
* History of seizures or epilepsy
* Current opioid use or in acute opioid withdrawal
* Abrupt discontinuation of alcohol, benzodiazepines, barbiturates, antiepileptic drugs
* History of glaucoma
* Uncontrolled hypertension
* Severe renal impairment and/or Chronic kidney disease stage III or GFR <60
* Acute hepatitis or liver failure
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis
* Use of antipsychotic medications or opiod analgesics
* Current or previous history of anorexia or bulimia nervosa
* Engagement with vomiting or laxative use within the last 28 days with the aim of controlling their shape or weight
* Current SSRI, SNRI, mood stabilizer, amphetamine, or corticosteroid use
* Current diagnosis of hyper or hypothyroidism or current use of thyroid replacement medicine
* Current use of beta blockers
* Current use of depo shot (medroxyprogesterone acetate) for birth control
* Current diagnosis of Cushing's disease or syndrome
* Current use of Monoamine Oxidase Inhibitors (MAOIs)
* Known hypersensitivity to bupropion, naltrexone, or metformin
* Any other reason rendering a participant unsuitable for trial participation, as determined by a clinician or study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent body weight change at 12 weeks | Baseline, 12 weeks
  Measurement of weight using a bluetooth body weight scale

SECONDARY OUTCOMES:
Change in body weight (in kg or pounds) at 12 weeks | Baseline, 12 weeks
  Measurement of weight using a bluetooth body weight scale
Physical Activity and Sedentary Behavior | Baseline, 12 weeks
  The Global Physical Activity Questionnaire (GPAQ) is a 16 item scale.
Dietary Intake | Baseline, 12 weeks
  Diet ID is powered by Diet Quality Photo Navigation (DQPN®). It is a digital toolkit and 1 component will be used in the study: ID assessment.
Habit/Automaticity | Baseline, 12 weeks
  The Self-Report Behavioral Automaticity Index (SRBAI) is a 4-item measure.
Hunger VAS (Visual Analogue Scale) | Baseline, 12 weeks
  The Hunger VAS (Visual Analogue Scale) is a reliable measure for appetite research. The Hunger VAS asks "How hungry did you feel over the past week" and is composed of a line with words anchored at each end describing the extremes (Not at all hungry, Extremely hungry). Participants are asked to make a mark on the line corresponding to their feelings and quantification of the measurement is done by measuring the distance from the left end of the mark.
Impact on Quality of Life | Baseline, 12 weeks
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life
Well-being | Baseline, 12 weeks
  The World Health Organization (WHO-5) Well-being Index consists of five statements, which respondents rate, in relation to the past two weeks, using a six-point Likert scale
Body Appreciation | Baseline, 12 weeks
  The Body Appreciation Scale (BAS-2) measures individuals acceptance of, favorable opinions toward, and respect for their bodies. There are 10 items, each assessed on a scale from 1-never to 5-always. Higher scores indicate higher body appreciation.
Self-Compassion | Baseline, 12 weeks
  The Self-Compassion Scale (SCS) is a 26-item measure of self-compassion that is psychometrically valid and theoretically coherent. The SCS consists of six subscales:
  self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identified.
  Subscales are computed by calculating the mean of subscale item responses. A total self-compassion score can be obtained by reverse scoring the negative subscale items (self-judgment, isolation, and over-identification) and computing a grand mean of all six subscale means. Higher scores indicate greater self compassion.
Weight Bias | Baseline, 12 weeks
  The Weight Bias Internalization Scale (WBIS-2F) has 13 items and responses are rated on a 7-point Likert scale(strongly disagree -strongly agree). Responses provide insight on the participant's internalized beliefs and feelings regarding their weight. There are two subscales: Weight-Related Distress (7 items; 7-13; Cronbach's alpha =0.910) and Weight-Related Self-Devaluation (6 items; 1-6; Cronbach's alpha =0.763). The WBIS-2F has been tested for validity in people with overweight and obesity and the two factor model demonstrated good to excellent fit with the data. Scores are calculated by taking an average of the response values. Questions 1,2,4,5, should be reverse scored before calculating the average. Higher scores indicating greater internalized weight bias.

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Alkhaddo, MD, Principal Investigator — WW International Inc
Locations (1):
- WW International, Inc, New York, New York, United States